CLINICAL TRIAL: NCT00272181
Title: A Phase II, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Proxinium in Patients With Advanced SCCHN Who Have Received at Least One Anti-Cancer Treatment Regimen for Advanced Disease
Brief Title: Study of Proxinium for Treating Patients With Squamous Cell Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual in North America
Sponsor: Sesen Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB4-845-01-IIA; NCT00335842 (obsolete NCT alias)
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms; Head and Neck Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Neoplasms, Squamous Cell; Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Determination (Experimental): The recommended dose (RD) for Proxinium is to be determined based on the rate of Dose Limiting Toxicities (DLT) within each dose cohort. The RD is to be established as the highest dose at which one or fewer patients out of six within a dose cohort experienced a DLT. The initial dose level is 500 μg of Proxinium in PBS (the amount of PBS used will be based on the estimated volume of the target tumour). Doses are to be escalated to a maximum of 700 μg or de-escalated to a minimum of 260 μg according to the prescribed algorithm outlined in the study protocol.
  Interventions: Drug: Proxinium

INTERVENTIONS:
Drug: Proxinium — Intratumoral administration of Proxinium directly to target tumors.

SUMMARY:
The purpose of this study is to determine the safety, effectiveness, and recommended dose of Proxinium in North American patients with Squamous Cell Head and Neck Cancer

DETAILED DESCRIPTION:
This study was an open-label, multicentre, dose determination study evaluating the safety and tolerability of Proxinium in the treatment of patients with advanced SCCHN who had received at least one anti-cancer treatment regimen for advanced disease. Fifteen patients were enrolled at nine sites. All patients with histologically confirmed SCCHN who had advanced disease were considered potential candidates for study entry.

Patients completed two phases of screening termed Initial Screening and Final Screening. Initial Screening assessed the EpCAM status of the patient's SCCHN prior to final screening procedures taking place. Patients had to have a biopsy of their advanced disease that had been appropriately collected for verification of EpCAM-positive SCCHN by immunohistochemical methods. If EpCAM-positive SCCHN was confirmed, the patient could enter Final Screening to determine full eligibility for participation in the study. At the beginning of Final Screening, all patients had to have received at least one anti-cancer treatment regimen for advanced disease. Patients who had successfully completed both Initial and Final Screening had a Principal Target Tumour and up to five additional Target Tumours designated for treatment prior to Day 1 dosing. Only one target tumour per week was to be injected. The Investigator was to treat the principal target tumour until clinically relevant tumour control of the principal target tumour was achieved, at which point other target tumours could be chosen and injected once per week at the same dose level of Proxinium.

The study was to comprise two stages. In Stage I, the recommended dose (RD) for Proxinium was to be determined based on the rate of dose-limiting toxicities (DLTs) within each dose cohort. A DLT was defined as the occurrence of excessive toxicity during the first four weeks of each patient's treatment with Proxinium during Stage I of the study, before the RD had been determined. The RD was to be established as the highest dose at which one or fewer patients out of six within a dose cohort experienced a DLT. The initial dose level was to be 500 µg, and three patients were to be initially enrolled into this dose cohort.

Doses were to be escalated to a maximum of 700 µg or de-escalated to a minimum of 260 µg according to the prescribed algorithm outlined in the study protocol and based on the number of patients experiencing a DLT within each dose cohort. Safety data was to be reviewed by the medical monitor, the site investigators who had enrolled patients at that dose, and Viventia Biotech Inc. (the sponsor) to determine if escalation or de-escalation was to occur. All Stage I patients, including those in the original RD cohort, were to remain in Stage I and continue treatment beyond their initial four weeks at their original dose assignment. If dose de-escalation was deemed necessary, all Investigators with patients receiving higher doses would have been notified and given the option of either administering a de-escalated dose or discontinuing treatment.

Stage II was to commence once the RD had been determined and an independent third party had reviewed the safety data. Patients enrolled subsequently were to receive treatment at the RD.

The RD cohort was to be expanded to include a total of 15 patients, and safety and efficacy evaluation was to continue being assessed.

Continued safety and tolerability as well as response rates, therapeutic endpoints, survival time, PK parameters, and immunogenicity were evaluated. Regardless of dose cohort, all patients were to be treated until complete resolution of all accessible Target Tumours, clinically relevant tumour progression, or until study drug suspension or withdrawal criteria had been met.

Four weeks after the end-of-treatment visit, patients were to return to the site for a follow-up visit that was to include a CT scan of the head and neck as well as other assessments, as described in the study protocol. Subsequently, patients were to enter the post-study surveillance period.

Enrolment in the study was halted before the RD of Proxinium was determined, and hence, Stage II of this study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

* Histologically confirmed recurrent squamous cell carcinoma of the head and neck.
* Immunohistochemically confirmed epithelial cell adhesion molecule (EpCAM)-positive SCCHN.
* Must have at least 1 accessible target tumor that is amenable to adequate direct injection.
* The patient must have at least 1 accessible target tumor without direct carotid artery involvement.

Prior/Concurrent Therapy:

* The patient must have received therapy for their primary disease
* The patient must have been diagnosed with persistent or recurrent disease or a second primary tumour.
* The patient's disease must be refractory.
* There must be at least 2 weeks between the last dose of chemotherapy or radiotherapy and receiving study drug or 4 weeks between the last dose of an experimental drug and receiving study drug.

Patient Characteristics:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Life expectancy of at least 12 weeks.
* Adequate hepatic function ALT and AST and total bilirubin levels ≤1.5 times ULN.
* Adequate renal function (serum creatinine <2.0 mg/dL).
* Hematologic values consisting of granulocytes ≥1500/μL, platelets ≥100 000/μL, and hemoglobin >8 g/dL.
* Prothrombin time and partial thromboplastin time within normal limits

Other:

* The patient must provide written informed consent.
* Fertile patients must use effective contraception

Exclusion Criteria:

* Brain tumor or brain metastases.
* Nasopharyngeal SCCHN.
* Human immunodeficiency virus, hepatitis C virus, or hepatitis B surface antigen.
* Uncontrolled bleeding from any target tumor(s) that are being considered for treatment or a history of tumor hemorrhage that has required medical intervention (other than direct compression).
* The patient is a candidate for surgical tumor resection of their target tumor(s).
* Pregnant or lactating.
* Clinically significant renal or hepatic disease.
* Requires regular use of aspirin, full-dose warfarin, or heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and recommended dose (RD) of Proxinium | Weekly dosing

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Cuthbert, Study Director — Sesen Bio, Inc.
Locations (19):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA Medical Center, Los Angeles, California
  - John P. Thropay, MD, Montebello, California
  - Mile High Oncology, Denver, Colorado
  - M.D. Anderson Cancer Center Orlando, Orlando, Florida
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Portland VA Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Mary Crowley Medical Research Center, Dallas, Texas
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUQ, L'Hotel-Dieu de Quebec, Québec, Quebec